CLINICAL TRIAL: NCT05716633
Title: Tracking the ENcapsulation of Pancreatic Collections in Acute Necrotizing Pancreatitis. A Serial MRI Based Prospective Study (MRI-ENCAP Study)
Brief Title: Tracking ENcapsulation of Pancreatic Collections in Acute Necrotizing Pancreatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Pankaj Gupta, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: 32055
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Acute Necrotizing Pancreatitis
Keywords: Acute Pancreatitis,Necrotic Collections,Walled off Necrosis
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Pancreatitis: Patients with acute pancreatitis will undergo serial MRI
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Serial MRI scans will be performed starting at day 15 from date of pain. Subsequent scans will be performed at 5 days interval till the clinically significant encapsulation (for all the collections in an individual patient) is seen.

SUMMARY:
The goal of this study is to investigate the encapsulation of fluid collections in patients with ANP using serial MRI.

The main questions it aims to answer are:

* Evaluating the timing of encapsulation of necrotic fluid collection using serial non-enhanced MRI.
* Identifying the factors that affect the timing of encapsulation of necrotic fluid collections Participants will undergo serial MRI scans (all with the same protocol) performed starting at day 15. Subsequent scans will be performed at 5 days interval till the clinically significant encapsulation (for all the collections in an individual patient) is seen or patients are excluded from the protocol due to intervention.

DETAILED DESCRIPTION:
Consecutive patients with ANP presenting to the hospital within 2 weeks from the pain onset will be recruited. They will undergo serial non-contrast MRI starting at day 15 and every 5 days thereafter, till complete encapsulation of PFC. Ultrasound evaluation of the collection will be performed on the day of MRI by a radiologist not involved in evaluation of MRI. The site and volume of collection as well as thickness and completeness of the capsule and solid content within the collection will be recorded independently by two radiologists. The timing of clinically significant (>50% of PFC show capsule) and complete encapsulation will be recorded. The proportion of collections encapsulating in each week after 2nd week of illness will be recorded. The association between timing of encapsulation and clinical/biochemical parameters will be assessed. The correlation between the degree of encapsulation and percentage of solid components will also be documented. Multivariate analysis will be performed to identify factors associated with timing of encapsulation.

ELIGIBILITY:
Inclusion Criteria:

1. Acute necrotizing pancreatitis
2. Presentation to hospital within 2 weeks of pain onset

2. Willing to give informed consent

Exclusion Criteria:

1. Contraindications to non- enhanced MRI (Claustrophobia, cardiac pacemaker, cochlear implant).
2. Acute on chronic pancreatitis
3. Mechanical ventilation, ionotropic support (precluding safe environment in MRI).
4. Drainage or aspiration of a collection prior to recruitment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with ANP presenting to the hospital within 2 weeks from the pain onset will be recruited. They will undergo serial non-contrast MRI starting at day 15 and every 5 days thereafter, till complete encapsulation of PFC. Ultrasound evaluation of the collection will be performed on the day of MRI by a radiologist not involved in evaluation of MRI.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Timing of Encapsulation | 1-2 months after initial MRI
  MRI scans will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Gupta, Principal Investigator — PGIMER, CHANDIGARH
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, Punjab, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baron TH, DiMaio CJ, Wang AY, Morgan KA. American Gastroenterological Association Clinical Practice Update: Management of Pancreatic Necrosis. Gastroenterology. 2020 Jan;158(1):67-75.e1. doi: 10.1053/j.gastro.2019.07.064. Epub 2019 Aug 31. PMID 31479658
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] ASGE Standards of Practice Committee; Muthusamy VR, Chandrasekhara V, Acosta RD, Bruining DH, Chathadi KV, Eloubeidi MA, Faulx AL, Fonkalsrud L, Gurudu SR, Khashab MA, Kothari S, Lightdale JR, Pasha SF, Saltzman JR, Shaukat A, Wang A, Yang J, Cash BD, DeWitt JM. The role of endoscopy in the diagnosis and treatment of inflammatory pancreatic fluid collections. Gastrointest Endosc. 2016 Mar;83(3):481-8. doi: 10.1016/j.gie.2015.11.027. Epub 2016 Jan 13. No abstract available. PMID 26796695
- [Background] Trikudanathan G, Tawfik P, Amateau SK, Munigala S, Arain M, Attam R, Beilman G, Flanagan S, Freeman ML, Mallery S. Early (<4 Weeks) Versus Standard (>/= 4 Weeks) Endoscopically Centered Step-Up Interventions for Necrotizing Pancreatitis. Am J Gastroenterol. 2018 Oct;113(10):1550-1558. doi: 10.1038/s41395-018-0232-3. Epub 2018 Oct 2. PMID 30279466
- [Background] Oblizajek N, Takahashi N, Agayeva S, Bazerbachi F, Chandrasekhara V, Levy M, Storm A, Baron T, Chari S, Gleeson FC, Pearson R, Petersen BT, Vege SS, Lennon R, Topazian M, Abu Dayyeh BK. Outcomes of early endoscopic intervention for pancreatic necrotic collections: a matched case-control study. Gastrointest Endosc. 2020 Jun;91(6):1303-1309. doi: 10.1016/j.gie.2020.01.017. Epub 2020 Jan 18. PMID 31958461
- [Background] van Grinsven J, van Brunschot S, van Baal MC, Besselink MG, Fockens P, van Goor H, van Santvoort HC, Bollen TL; Dutch Pancreatitis Study Group. Natural History of Gas Configurations and Encapsulation in Necrotic Collections During Necrotizing Pancreatitis. J Gastrointest Surg. 2018 Sep;22(9):1557-1564. doi: 10.1007/s11605-018-3792-z. Epub 2018 May 11. PMID 29752684
- [Background] Chantarojanasiri T, Yamamoto N, Nakai Y, Saito T, Saito K, Hakuta R, Ishigaki K, Takeda T, Uchino R, Takahara N, Mizuno S, Kogure H, Matsubara S, Tada M, Isayama H, Koike K. Comparison of early and delayed EUS-guided drainage of pancreatic fluid collection. Endosc Int Open. 2018 Dec;6(12):E1398-E1405. doi: 10.1055/a-0751-2698. Epub 2018 Nov 23. PMID 30505932
- [Background] Rana SS, Sharma R, Kishore K, Dhalaria L, Gupta R. Safety and Efficacy of Early (<4 Weeks of Illness) Endoscopic Transmural Drainage of Post-acute Pancreatic Necrosis Predominantly Located in the Body of the Pancreas. J Gastrointest Surg. 2021 Sep;25(9):2328-2335. doi: 10.1007/s11605-021-04945-y. Epub 2021 Feb 5. PMID 33547585
- [Background] Rana SS, Verma S, Kang M, Gorsi U, Sharma R, Gupta R. Comparison of endoscopic versus percutaneous drainage of symptomatic pancreatic necrosis in the early (< 4 weeks) phase of illness. Endosc Ultrasound. 2020 Nov-Dec;9(6):402-409. doi: 10.4103/eus.eus_65_20. PMID 33318376